CLINICAL TRIAL: NCT00523289
Title: Cardiovascular Safety Research: Bupivacaine With Vasoconstrictor Versus Ropivacaine in Brachial Plexus Block
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Sao Paulo (Other)
Collaborators: Cristália Produtos Químicos Farmacêuticos Ltda. (Industry)
Responsible Party: José O.Costa Auler Jr - Full prof.Anesthesiology USP, University Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: CRT029
Record Dates: First submitted 2007-08-29; First posted 2007-08-31 (Estimated); Last update posted 2009-02-19 (Estimated); Status verified 2009-02

CONDITIONS: Injuries, Hand; Anesthesia Conduction; Anesthetics, Local
Keywords: Ropivacaine; Bupivacaine; Upper Extremity; Local anesthetic
MeSH Terms: conditions — Hand Injuries | interventions — Bupivacaine; Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- B (Active Comparator): Arm number B corresponds to the Bupivacaine group.
  Interventions: Drug: Bupivacaine
- R (Active Comparator): Arm number R corresponds to the Ropivacaine group.
  Interventions: Drug: Ropivacaine

INTERVENTIONS:
Drug: Bupivacaine — Dosage: 150mg at once for anesthesia induction
  Arms: B
Drug: Ropivacaine — Single dose of ropivacaine, 150mg
  Arms: R

SUMMARY:
The purpose of this study is to determine if bupivacaine (75% levobupivacaine plus 25% racemic bupivacaine) with vasoconstrictor is effective and safety as ropivacaine in brachial plexus block for orthopedic surgery.

DETAILED DESCRIPTION:
The intoxication by Bupivacaine is considered life threatening. Currently the most safety local anesthetic in substitution to bupivacaine is ropivacaine, however in Brasil there is a bupivacaine mixture of 75% levobupivacaine plus 25% racemic bupivacaine. The research design is:

Patients involved: 48; age: 18 to 40 years old; both sex; ASA I and II. Surgery: elective upper extremity orthopedic surgery. Anesthesia technique: brachial plexus block. Primary endpoint: cardiovascular safety; analysis by continuous Holter. Secondary endpoint: anesthetic and analgesic efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Patients involved: 48; ASA I and II;
* Surgery: elective upper extremity orthopedic surgery.

Exclusion Criteria:

* Contraindications to anesthesia technique and/or to local anesthetic;
* Participation in different trials in the last two months;
* Antiretroviral users;
* Obesity.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2007-10; Primary Completion 2009-03 (Estimated); Study Completion 2009-07 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular safety | Two days

SECONDARY OUTCOMES:
Anesthesia Analgesia quality | Two days

CONTACTS AND LOCATIONS:
Overall Officials: José Otávio C Auler Junior, PhD/Chairman, Study Chair — Hospital das Clínicas - Medicine School of the University of São Paulo

REFERENCES:
- [Background] Casati A, Santorsola R, Aldegheri G, Ravasi F, Fanelli G, Berti M, Fraschini G, Torri G. Intraoperative epidural anesthesia and postoperative analgesia with levobupivacaine for major orthopedic surgery: a double-blind, randomized comparison of racemic bupivacaine and ropivacaine. J Clin Anesth. 2003 Mar;15(2):126-31. doi: 10.1016/s0952-8180(02)00513-5. PMID 12719052
- [Background] Casati A, Chelly JE, Cerchierini E, Santorsola R, Nobili F, Grispigni C, Di Benedetto P, Torri G. Clinical properties of levobupivacaine or racemic bupivacaine for sciatic nerve block. J Clin Anesth. 2002 Mar;14(2):111-4. doi: 10.1016/s0952-8180(01)00364-6. PMID 11943523
- [Background] Casati A, Borghi B, Fanelli G, Montone N, Rotini R, Fraschini G, Vinciguerra F, Torri G, Chelly J. Interscalene brachial plexus anesthesia and analgesia for open shoulder surgery: a randomized, double-blinded comparison between levobupivacaine and ropivacaine. Anesth Analg. 2003 Jan;96(1):253-9, table of contents. doi: 10.1097/00000539-200301000-00051. PMID 12505962
- [Background] Santorsola R, Casati A, Cerchierini E, Moizo E, Fanelli G. [Levobupivacaine for peripheral blocks of the lower limb: a clinical comparison with bupivacaine and ropivacaine]. Minerva Anestesiol. 2001 Sep;67(9 Suppl 1):33-6. Italian. PMID 11778092
- [Background] Borgeat A, Ekatodramis G, Blumenthal S. Interscalene brachial plexus anesthesia with ropivacaine 5 mg/mL and bupivacaine 5 mg/mL: effects on electrocardiogram. Reg Anesth Pain Med. 2004 Nov-Dec;29(6):557-63. doi: 10.1016/j.rapm.2004.09.005. PMID 15635515